CLINICAL TRIAL: NCT00564356
Title: The Safety of Cataract Removal by Phacoemulsification Surgery in Patients Under Anti-aggregant and Coumadin Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sheba Medical Center, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-07-3017-OS-CTIL
Record Dates: First submitted 2007-11-26; First posted 2007-11-27 (Estimated); Last update posted 2009-07-21 (Estimated); Status verified 2009-07

CONDITIONS: Efficacy; Complications
Keywords: cataract, phacoemulsification, coumadin, antiaggregants
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction; Phacoemulsification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Other): patients under coumadin and antiaggregants operated by phacoemulsification
  Interventions: Procedure: cataract surgery with phacoemulsification

INTERVENTIONS:
Procedure: cataract surgery with phacoemulsification — removal of cataract with phacoemulsification technique

SUMMARY:
To assess the risks of intra- and postoperative bleeding tendency associated with cataract surgery by phacoemulsification in patients on coumadin and antiaggregant treatments.

Design: Consecutive prospective study.

DETAILED DESCRIPTION:
To assess the risks of intra- and postoperative bleeding tendency associated with cataract surgery by phacoemulsification technique in patients on coumadin and antiaggregant treatment Design: Consecutive prospective study.

ELIGIBILITY:
Inclusion Criteria:

* patients who give informed consent to participate in the study

Exclusion Criteria:

* single eye complicated cataract

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-08 (Actual); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
safety and efficacy of cataract surgery with phacoemulsification under coumadin and antiaggregant treatment | 3.5 years

SECONDARY OUTCOMES:
other complications | 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ophira Salomon, Study Director — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Result] Barequet IS, Sachs D, Priel A, Wasserzug Y, Martinowitz U, Moisseiev J, Salomon O. Phacoemulsification of cataract in patients receiving Coumadin therapy: ocular and hematologic risk assessment. Am J Ophthalmol. 2007 Nov;144(5):719-723. doi: 10.1016/j.ajo.2007.07.029. Epub 2007 Sep 17. PMID 17870045